CLINICAL TRIAL: NCT06174441
Title: The Effect of 24-week Dietary Intake of Food Supplements on Hair: Double Blind, Placebo-controlled, Randomised Three-way Study to Assess Effectiveness of Two Test Products
Brief Title: The Effect of 24-week Dietary Intake of Food Supplements on Hair
Acronym: TO-HAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIST - Faculty of Applied Sciences (Other)
Collaborators: Slovenian Research and Innovation Agency (Unknown); Tosla d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIST TO-HAIR 01-2023
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2023-12

CONDITIONS: Hair Thinning; Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1 (CPMSM) (Active Comparator): Investigational product 1: daily dose 25 mL contains: Hydrolyzed fish collagen 5 g, methylsulphonylmethane (MSM) 1,5 g, Biotin 150 μg, Vitamin B6 1,6 mg, Zinc 2 mg, Vitamin C 120 mg.
  Interventions: Dietary Supplement: Investigational product 1 (CPMSM)
- Test group 2 (HC+) (Active Comparator): Investigational product 2: daily dose 25 mL contains: Niacin 16 mg, Pantothenic acid 6 mg, Biotin 500 μg, Vitamin B6 1,4 mg, Folic acid 200 μg, Zinc 2 mg, Pea sprout extract 100 mg, Horsetail aerial parts extract 70 mg, Ashwagandha root extract 40 mg, Saw palmetto fruit extract 40 mg, Nettle leaves extract 30 mg, Grape seed extract 10 mg.
  Intervention: Dietary Supplement: Placebo Placebo group (PG) will receive placebo product without any of the active ingredients (PL, daily dose 25 mL: no active ingredients).
  Interventions: Dietary Supplement: Investigational product 2 (HC+)
- Placebo group (Placebo Comparator): placebo product without any of the active ingredients, daily dose 25 mL: no active ingredients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Investigational product 1 (CPMSM) — Test group 1 will receive investigational product 1 (CPMSM: daily dose 25 mL contains: Hydrolyzed fish collagen 5 g, methylsulphonylmethane (MSM) 1,5 g, Biotin 150 μg, Vitamin B6 1,6 mg, Zinc 2 mg, Vitamin C 120 mg).
  Arms: Test group 1 (CPMSM)
Dietary Supplement: Investigational product 2 (HC+) — Test group 2 (TG2) will receive investigational product 2 (HC+: daily dose 25 mL contains: Niacin 16 mg, Pantothenic acid 6 mg, Biotin 500 μg, Vitamin B6 1,4 mg, Folic acid 200 μg, Zinc 2 mg, Pea sprout extract 100 mg, Horsetail aerial parts extract 70 mg, Ashwagandha root extract 40 mg, Saw palmetto fruit extract 40 mg, Nettle leaves extract 30 mg, Grape seed extract 10 mg).
  Arms: Test group 2 (HC+)
Dietary Supplement: Placebo — Placebo group (PG) will receive placebo product without any of the active ingredients (PL, daily dose 25 mL: no active ingredients).
  Arms: Placebo group

SUMMARY:
Purpose of this randomized, double-blind, placebo-controlled study will be to evaluate whether the daily use of novel dietary supplements over 24 weeks is able strengthen and promote growth of hairs, improve their density and thickness and reduce hair loss in adults with self-perceived thinning hair.

DETAILED DESCRIPTION:
Single centre, randomized, double-blind, placebo-controlled, one-period effectiveness study to evaluate whether the daily use of novel dietary supplements over 24 weeks will strengthen and promote density and quality of hair in adults with self-perceived thinning hair.

Study population will be divided in three groups - 32 in active groups and 20 in placebo group. Test group 1 (TG1) will receive investigational product 1 (CPMSM: containing fish collagen, methylsulphonylmethane (MSM), vitamins and zinc), test group 2 (TG2) will receive investigational product 2 (HC+: containing mixture of herbal extracts, B-vitamins and zinc) and the placebo group (PG) will receive placebo product without any of the active ingredients (PL, no active ingredients). Participants will test continuous administration of placebo or investigational products (in the form of syrups) for 24 weeks in order to demonstrate and assess multiple-dose effects.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian volunteers of both sexes; aged 25-60 years at the time of the signature of Informed consent form (ICF).
* Darker (not blonde or grey) at least 5 cm long on midline.
* Signed Informed consent form (ICF).
* Fitzpatrick skin phototypes I-IV.
* Self-perceived hair thinning - subjects complaining of hair fall and damage.
* Derived Sinclair Scale score up to 3.
* In good general health condition.
* Subjects who are not crash dieting.
* Willingness to maintain using regular hair care routine regarding hair washing and styling, hair dye / hair colour during the study period.
* Willingness to refrain from any type of hair treatment like perming, permanent straightening etc. during the study duration.
* Willingness to not substantially change their lifestyle, current diet, medications, or exercise routines for the duration of the study.
* Willingness to refrain from any other topical treatment/hair spa and oral medications or supplement for hair growth during the study.
* BMI < 35
* Willingness to avoid a consumption of any other food supplements containing methylsulfonylmethane (MSM), antioxidants, collagen or other protein-based food supplements, Pea sprout extract, Horsetail extract, Ashwagandha root extract, Saw palmetto fruit extract, Nettle leaves extract, Grape seed extract, biotin, zinc, niacin, pantothenic acid, vitamin B6, folic acid during the study.
* Willingness to follow all study procedures and keeping a diary during the study (to follow their compliance and palatability).
* Willingness not to begin or change any estrogen or progesterone or other hormonal therapies.
* Willingness of subjects who have color treated hair to have the color treatment performed at the same time interval prior to each visit.
* No known or suspected allergy to any ingredient of the tested products as established by medical history.

Exclusion Criteria:

* Pregnancy or breastfeeding or planning pregnancy in near future (in next year).
* Menopausal female subjects as determined by medical history.
* Recent initiation or change (<6 months) of hormones for birth control or hormone replacement therapy in females or other hormonal therapies.
* Use of treatments for hair growth treatment including minoxidil, finasteride or light therapy within the last 3 months or other medications that are known to cause hair loss or affect hair growth (eg. Cyproterone acetate, Aldactone/spironolactone, 5-alpha-reductase inhibitors, phenytoin) within the last 6 months.
* Subjects with any clinically significant history of underlying uncontrolled medical illness including thyroid disorders, diabetes mellitus, hypertension, cancer, HIV, hepatitis, severe anemia, serious disorder of heart and respiratory apparatus or any other serious medical illness.
* Changes in dietary habits and dietary supplementation in the last three months prior to inclusion.
* Veganism.
* Regular use of food supplements containing methylsulfonylmethane (MSM), collagen or other protein-based food supplements, Pea sprout extract, Horsetail extract, Ashwagandha root extract, Saw palmetto fruit extract, Nettle leaves extract, Grape seed extract, or vitamin or antioxidant supplements, which will compromise the study, in the last three months prior to inclusion.
* Subjects having any active scalp or skin disease which may interfere with the study treatment and evaluations.
* Subjects who have had hair transplant.
* Subjects undergoing any chemical hair salon treatment-straightening / perming.
* Subjects participating in other similar cosmetic or therapeutic trial within last year.
* Subjects who have experienced a known stressful event within the last 6 months such as death in family, miscarriage etc.
* Known history or recent blood work indicating iron deficiency, bleeding disorders or platelet dysfunction syndrome.
* Smokers with usage > 20 cigarettes/day.
* Changes in hair care routine in the last month prior to inclusion,
* Mental incapacity that precludes adequate understanding or cooperation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Change of hair density from baseline in all test groups in comparison to placebo group after 24 weeks of dietary supplementation | 24-weeks
  Significant change of hair density from baseline in test groups, in comparison to placebo group after 24 weeks of dietary supplementation with study products is expected. Hair density will be assessed through trichoscopy using H2H matching procedure. Results will be analysed for whole sample and separately for men and women.

SECONDARY OUTCOMES:
Change of scalp sebum from baseline in all test groups in comparison to placebo group after 24 weeks of dietary supplementation | 24 weeks
  Significant change of scalp sebum from baseline in test groups, in comparison to placebo group after 24 weeks of dietary supplementation with study products is expected. Scalp sebum will be measured using DermaLab SkinLab sebum module.
Change of hair thickness from baseline in all test groups in comparison to placebo group after 24 weeks of dietary supplementation | 24-weeks
  Significant change of hair thickness from baseline in test groups, in comparison to placebo group after 24 weeks of dietary supplementation with study products is expected. Hair thickness will be assessed through trichoscopy using H2H matching procedure and average hair thickness determined.
Change of hair loss from baseline in all test groups in comparison to placebo group after 24 weeks of dietary supplementation | 24-weeks
  Significant change of hair loss from baseline in test groups, in comparison to placebo group after 24 weeks of dietary supplementation with study products is expected. Hair loss will be assessed through Hair comb test.
Change of terminal hair density from baseline in all test groups in comparison to placebo group after 24 weeks of dietary supplementation | 24 weeks
  Significant change of hair density from baseline in test groups, in comparison to placebo group after 24 weeks of dietary supplementation with study products is expected. Hair density will be assessed through trichoscopy using H2H matching procedure. Results will be analysed for whole sample and separately for men and women.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Žmitek, PhD, Study Director — Head of research group
Locations (1):
- VIST - Faculty of Applied Sciences, Institute of Cosmetics, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No